CLINICAL TRIAL: NCT06281236
Title: A Trial of Prednisolone in Combination With SPI-62 in Participants With Polymyalgia Rheumatica (PMR)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: lack of enrollment
Sponsor: Sparrow Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SPI-62-CL-1002
Record Dates: First submitted 2024-02-20; First posted 2024-02-28 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Polymyalgia Rheumatica
MeSH Terms: conditions — Polymyalgia Rheumatica | interventions — Prednisolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- prednisolone + SPI-62 (Experimental): Participants will receive prednisolone throughout the trial and SPI-62 on days 3-16.
  Interventions: Drug: Prednisolone; Drug: SPI-62

INTERVENTIONS:
Drug: Prednisolone — Prednisolone according to the participant's pre-trial dose, symptoms and inflammatory biomarkers.
Drug: SPI-62 — SPI-62 administered once daily.

SUMMARY:
This will be an open label phase 1b trial to characterize the pharmacodynamics and PK of prednisolone and SPI-62 when co-administered to participants with PMR. Up to 24 participants could be recruited.

DETAILED DESCRIPTION:
This will be an open label phase 1b trial to characterize the pharmacodynamics and PK of prednisolone and SPI-62 when co-administered to participants with PMR. Up to 24 participants could be recruited.

Patients diagnosed with PMR whose PMR symptoms do not vary in intensity or frequency to the degree that a clinically indicated increase in prednisolone prescription might be anticipated will be included in the trial.

Participants will continue to receive prednisolone and will receive SPI-62 from Days 3-16

Inflammatory biomarkers, symptom measures, biomarkers of prednisolone toxicity, PK of prednisolone and SPI-62, and biomarkers of SPI-62 pharmacological activity will be measured on Days 2, 3, and 16. ABPM will be monitored on days 1 and 15.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Diagnosis of PMR according to European League Against Rheumatism and American College of Rheumatology classification criteria confirmed by a rheumatologist
* Absence of PMR relapse based on symptoms and acute phase markers
* Daily oral prednisolone 10, 12.5, 15, 17.5, or 20 mg dose that will have been stable for at least 7 days prior to Day 1

Exclusion Criteria:

* Any contraindication for prednisolone administration
* A diagnosis or any clinical features of giant cell arteritis
* Any autoimmune disease (e.g., late-onset rheumatoid arthritis) other than PMR
* Use of medications for treatment of PMR other than oral prednisolone within specified intervals prior to Day 1 and during the treatment period
* Use of other medications likely to interfere with trial assessments
* History or diagnosis of endogenous hypercortisolism
* Any current or prior medical condition, medical or surgical therapies, or clinical trial participation expected to interfere with the conduct of the trial or the evaluation of its results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2022-02-22 (Actual); Primary Completion 2025-03-25 (Actual); Study Completion 2025-04-25 (Actual)

PRIMARY OUTCOMES:
Erythrocyte sedimentation rate | Baseline to Day 28
C-reactive protein | Baseline to Day 28
Plasma fibrinogen | Baseline to Day 28

CONTACTS AND LOCATIONS:
Overall Officials: David Katz, Study Chair — Sparrow Pharmaceuticals
Locations (5):
- Germany (5):
  - Emovis Gmbh, Berlin
  - Klinische Forschung Hannover Mitte GmbH/Pratia, Hanover
  - Universitätsmedizin der Johannes Gutenburg Universität Mainz, Mainz
  - Klinikum der Universität München, München
  - Klinische Forschung Schwerin GmbH/Pratia, Schwerin

IPD SHARING:
Plan to Share IPD: No